CLINICAL TRIAL: NCT04533958
Title: Evaluation of Hypnosis in Virtual Reality on the Anxiety of Patients With Metastatic Prostate Cancer Over Chemotherapy Monocentric, Comparative, Randomized, Open Study
Brief Title: Evaluation of Hypnosis in Virtual Reality on the Anxiety of Patients With Metastatic Prostate Cancer Over Chemotherapy
Acronym: HypProMet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Gregoire Private Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-A03336-51
Record Dates: First submitted 2020-08-11; First posted 2020-09-01 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Prostate Cancer
Keywords: Virtual reality; Oncology; Chemotherapy; Anxiety
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HypnoVR Arm (Experimental): During each Docetaxel infusion, patients benefit from a 20-minute session of medical hypnosis in virtual reality.
  Interventions: Device: HYPNO VR® device
- Control Arm (No Intervention): Patients receive the docetaxel infusions under standard conditions (no medical hypnosis in virtual reality intervention)

INTERVENTIONS:
Device: HYPNO VR® device — The HYPNO VR® device is a software application of medical hypnosis in the treatment of pain and anxiety. It is associated with equipment: a virtual reality headset and a headphone.
  Before each Docetaxel infusion, the nursing staff offers patients the choices: visual universe, musical theme, male or female voice. The nursing staff selects the chemotherapy program, selects a duration of 20 minutes and presses start to start the medical hypnosis session in virtual reality.
  After completing the hypnotic trance sequence, as in a classic session, the patient is brought back to the "return" and exit hypnosis phase under the supervision of the nursing staff.
  Arms: HypnoVR Arm

SUMMARY:
Prostate cancer is the first cancer in men. The treatment of metastatic prostate cancer with chemotherapy is based on the intravenous administration of docetaxel chemotherapy. Symptoms of anticipatory nausea, linked to anxiety caused by the treatment, may occur. Hypnosis is already used to treat the anxiety of people with cancer and can help treat the symtoms of nausea and vomiting of women with breast cancer.

The purpose of the study is to evaluate the effect of medical hypnosis in virtual reality on the anxiety of patients with metastatic prostate cancer receiving Docetaxel chemotherapy treatment in comparison with a control group.

DETAILED DESCRIPTION:
After verifying the patient's eligibility criteria and obtaining the signed informed consent form, the patient is randomized to the arm receiving hypnosis in virtual reality or to the control arm. The study ends after the 12 courses of docetaxel or premature termination of the study.

ELIGIBILITY:
Inclusion Criteria:

* Man aged ≥ 18 years
* Histologically proven metastatic prostate adenocarcinoma,
* Patient undergoing chemotherapy according to the following conventional scheme: 12 courses of Docetaxel every two weeks
* Patient who signed their informed consent
* Patient benefiting from social security coverage
* Patient treated and followed in the center for the duration of the study (6 months maximum).

Exclusion Criteria:

* Patient participating in another clinical trial on an experimental molecule
* Patient who received previous chemotherapy
* Patient unable to submit to protocol monitoring for psychological, social, family or geographic reasons
* Patient deprived of their liberty or under guardianship
* Patient with underlying or concomitant pathology incompatible with inclusion in the trial, whether psychiatric or somatic

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Demonstrate a modification in anxiety after each infusion of Docetaxel in the HypnoVR arm compared to the control arm. | For up to 6 months, every 2 weeks (before and after the 12 infusions), starting on day of first infusion until day of the last twelfth infusion
  Comparison of anxiety by the State Trait Anxiety Inventory (STAI) score before and after each docetaxel infusion (i.e. 24 questionnaires) between the HypnoVR arm and the control arm. The score is a quantitative variable with values ranging from 20 to 80. The higher the score is, the more important the anxiety is.

SECONDARY OUTCOMES:
Test the hypothesis that medical hypnosis in virtual reality is accompanied by a decrease in nausea before and after the Docetaxel cures | For up to 6 months, every 2 weeks (before and after the 12 infusions), starting on day of first infusion until day of the last twelfth infusion
  Comparison of nausea (Analogical Visual Scale-VAS) before and after each infusion and at the end of treatment (i.e. 24 questionnaires) between the two arms. The analogical visual scale of nausea is a 6-point scale from "no nausea" to "maximum nausea". The higher the score is, the more important nausea are.
Test the hypothesis that medical hypnosis in virtual reality is accompanied by a decrease in vomiting before and after the Docetaxel cures | For up to 6 months, every 2 weeks (before and after the 12 infusions), starting on day of first infusion until day of the last twelfth infusion
  Comparison of the number of vomiting episodes (n) before and after each infusion and at the end of treatment (i.e. 24 questionnaires) between the two arms.
Test the hypothesis that medical hypnosis in virtual reality is accompanied by an increase in the quality of life by the EQ-5D-3L questionnaire for the health state description part after the end of treatment | For up to 6 months, one assessment questionnaire on day of inclusion and one assessment questionnaire at the end of study visit (month 6)
  Comparison of the quality of life by the EQ-5D-3L questionnaire before the start of treatment with Docetaxel and after the end of treatment (after 12 infusions, ie two questionnaires) between the two arms. The EQ-5D-3L questionnaire has two components: health state description and evaluation. In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The respondents self-rate their level of severity for each dimension using three-level (EQ-5D-3L).
Test the hypothesis that medical hypnosis in virtual reality is accompanied by an increase in the quality of life by the EQ-5D-3L questionnaire for the health state evaluation part after the end of treatment | For up to 6 months, one assessment questionnaire on day of inclusion and one assessment questionnaire at the end of study visit (month 6)
  Comparison of the quality of life by the EQ-5D-3L questionnaire before the start of treatment with Docetaxel and after the end of treatment (after 12 infusions, ie two questionnaires) between the two arms. The EQ-5D-3L questionnaire has two components: health state description and evaluation. In the evaluation part, the respondents evaluate their overall health status using the visual analogic scale (EQ-VAS) from 0 (the worst state of health imaginable) to 100 (the best state of health imaginable).
Test the hypothesis that medical hypnosis in virtual reality is accompanied by an increase in the quality of life by the FACT-P (Functional Assessment of Cancer Therapy-Prostate) questionnaire after the end of treatment | For up to 6 months, one assessment questionnaire on day of inclusion and one assessment questionnaire at the end of study visit (month 6)
  Comparison of the quality of life by the FACT-P questionnaire before the start of treatment with Docetaxel and after the end of treatment (after 12 infusions, ie two questionnaires) between the two arms. The FACT-P is a multidimensional, self-report quality of life instrument specifically designed for use with prostate cancer patients. It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being, which is further supplemented by 12 site specific items to assess for prostate related symptoms. The respondents self-rate their level of severity for each item on a 5-points scale from 0 (not at all) to 4 (very much).
Test the hypothesis that medical hypnosis in virtual reality is accompanied by a good patient satisfaction after each infusion of Docetaxel | For up to 6 months, every 2 weeks (after each infusion), starting on day of first infusion until day of the last twelfth infusion (month 6)
  Evaluation of patient satisfaction in the HYPNO VR group by the patient self-questionnaire after each infusion of Docetaxel, i.e. 12 questionnaires. a level of satisfaction (on a 11-point scale from 0 to 10) of the patient will be measure for the state of relaxation, security, understanding, overall satisfaction.
Test the hypothesis that medical hypnosis in virtual reality is accompanied by a modification in the prescription of antiemetic treatments | For up to 6 months, every 2 weeks (before each infusion), starting on day of the first infusion until the day of the last twelfth infusion
  Comparison of the proportion of antiemetic treatment prescriptions (dosage/posology stopped, added or changed) for each course between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier ARTIGNAN, MD, Principal Investigator — CHP Saint Grégoire
Locations (6):
- France (3):
  - Clinique Pasteur-Lanroze, Brest
  - CHP Saint-Grégoire, Saint-Grégoire
  - Clinique de la Côte d'Emeraude, St-Malo
- Portugal (3):
  - Hospital Lusiadas Amadora, Amadora
  - Hospital Lusiadas Lisboa, Lisbon
  - Hospital Lusiadas Porto, Porto

IPD SHARING:
Plan to Share IPD: No